CLINICAL TRIAL: NCT00918775
Title: A Phase II Metastasectomy Study for Patients With Renal Cell Carcinoma
Brief Title: Follow-up After Metastasectomy in Patients With Kidney Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: 2009-0038; NCI-2017-00524 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2009-0038 (Other: M D Anderson Cancer Center); R01CA90370 (Other: National Cancer Institute)
Record Dates: First submitted 2009-06-10; First posted 2009-06-11 (Estimated); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Aftercare

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Observational (follow-up) (Other): After metastasectomy, patients are followed up every 6 months for up to 5 years.
  Interventions: Other: Follow-Up Care; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Other: Follow-Up Care — Undergo follow-up
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase II trial studies the follow-up after metastasectomy in patients with kidney cancer. Following up patients' health condition after metastasectomy may help doctors to learn if the surgical removal of the primary tumor or the parts of the cancer that has spread to other parts of the body is a good method for treating patients who have kidney cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the 24-week progression free/relapse free survival rate in patients undergoing metastasectomy for metastatic renal cell carcinoma (mRCC).

SECONDARY OBJECTIVES:

I. To evaluate progression free survival (PFS), relapse free survival (RFS) and overall survival (OS) in patients undergoing metastasectomy.

II. To evaluate tissue determinants predictive for resectability, PFS and OS in patients undergoing metastasectomy.

OUTLINE:

After metastasectomy, patients are followed up every 6 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically confirmed renal cell carcinoma (RCC)
* Patients have clinical reasons for undergoing a surgical resection of tumor; there are two main categories of patients:

  * Patients with fully resectable disease as defined by lesions accessible by a surgeon during no more than two separate surgical sessions, and are expected to be rendered surgically no evidence of disease (NED)
  * Patients undergoing a noncurative procedure for relief of symptoms or for management of threatening lesions
* Patients have been deemed resectable by the subspecialty surgeon involved in the patient's care
* Patients must give written informed consent prior to initiation of therapy, in keeping with the policies of the institution; patients with a history of major psychiatric illness must be judged able to fully understand the investigational nature of the study and the risks associated with the therapy; the only approved consent is attached to this protocol
* Patients must have ability to comply with study and/or follow-up procedures
* Members of all races and ethnic groups are eligible for this trial

Exclusion Criteria:

* Patients must not have active acute infections that could be worsened by surgery or interfere with this study
* Patients must not have clinically significant cardiovascular disease, or peripheral vascular disease that creates an unacceptably high operative risk
* Patients must not have history of other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates surgical resection, or render the subject at high risk from treatment complications
* Patients must not have a history of uncontrolled severe depression

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2009-06-09 (Actual); Primary Completion 2026-12-20 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
Binary indicator that the patient is alive with no evidence of disease progression (either progression or relapse) post surgery | 24 weeks
  Assessed using a logistic regression model.

SECONDARY OUTCOMES:
Progression free survival (PFS) | Up to 5 years
Overall survival (OS) | Up to 5 years
  Will be analyzed by Kaplan Meier plots and appropriate regression analyses using the vector of intervention indicators (ZD, ZE, ZI) as covariates, with the model determined by preliminary goodness-of-fit analyses.
Disease free survival (DFS) | Up to 5 years
  Will be analyzed by Kaplan Meier plots and appropriate regression analyses using the vector of intervention indicators (ZD, ZE, ZI) as covariates, with the model determined by preliminary goodness-of-fit analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Jonasch, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org